CLINICAL TRIAL: NCT02413645
Title: A Phase I, Open Label Dose Escalation Study to Evaluate Safety of iHIVARNA-01 in Chronically HIV-infected Patients Under Stable Combined Antiretroviral Therapy
Brief Title: Phase I, Open Label Dose Escalation Study to Evaluate Safety of iHIVARNA-01 in Chronically HIV-infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Judit Pich Martínez (Other)
Responsible Party: Sponsor-Investigator, Judit Pich Martínez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: iHIVARNA; 2014-004591-32 (EudraCT Number)
Record Dates: First submitted 2015-03-30; First posted 2015-04-10 (Estimated); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: HIV-infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — RNA, Messenger

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 100 μg TriMix mRNA (TriMix_100) (Other): Cohort 1 (control group) 3 patients will receive 100 μg of mRNA (i.e. 100 μg TriMix mRNA).If two or more of the three patients have a dose limiting toxicity (DLT), DSMB should be consulted and study will be terminated. If one or no patients have a dose limiting toxicity, three patients will be enrolled at the next dose level.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  Interventions: Biological: TriMix_100
- 300 μg TriMix mRNA (TriMix_300) (Other): Cohort 2 (control group) 3 patients will receive 300 μg of mRNA (i.e. 100 μg TriMix mRNA).If two or more of the three patients have a DLT, DSMB should be consulted and study will be terminated. If one or no patients have a dose limiting toxicity, three patients will be enrolled at the next dose level.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  Interventions: Biological: TriMix_300
- 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) (Experimental): Cohort 3 (experimental group) 3 patients will receive 600 μg of mRNA (300 μg HIV mRNA + 300 μg TriMix mRNA). If two or more of the three patients have a DLT, DSMB should be consulted and study will be terminated. If one or no patients have a dose limiting toxicity, three patients will be enrolled at the next dose level.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  Interventions: Biological: 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA)
- 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) (Experimental): Cohort 4 (experimental group) 3 patients will receive 900 μg of mRNA (i.e. 600 μg HIV mRNA and 300 μg TriMix mRNA). If two or more of the three first patients have a DLT, then additional three patients will be enrolled at the previous level dose (dose will be reduced to 600 μg of mRNA per vaccination). If one or no patients have a DLT, additional three patients will be enrolled at 900 μg dose level. If two or more of the six patients receiving 900 μg of mRNA have a DLT, then additional 3 patients will be enrolled at the previous level dose (dose will be reduced to 600 μg of mRNA per vaccination). If one or no patients of the six patients have a DLT, six patients will be enrolled at the next dose level.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  Interventions: Biological: 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA)
- 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA) (Experimental): Cohort 5 (experimental group) 6 patients will receive 1200 μg of mRNA (i.e. 900 μg HIV mRNA + 300 μg TriMix mRNA) in case one or no patients of the six patients at the previous dose level have a DLT.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  Interventions: Biological: 1200μg mRNA (900 μg HIV mRNA+300 μg TriMix mRNA)

INTERVENTIONS:
Biological: TriMix_100 — 100 μg of TriMix in
  Arms: 100 μg TriMix mRNA (TriMix_100)
Biological: TriMix_300 — 300 μg of TriMix in
  Arms: 300 μg TriMix mRNA (TriMix_300)
Biological: 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) — 600 μg of mRNA (300 μg TriMix + 300 μg HIVACAT)
  Other Names: iHIVARNA-01.1
  Arms: 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA)
Biological: 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) — 900 μg of mRNA (300 μg TriMix + 600 μg HIVACAT)
  Other Names: iHIVARNA-01.2
  Arms: 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA)
Biological: 1200μg mRNA (900 μg HIV mRNA+300 μg TriMix mRNA) — 1200 μg of mRNA (300 μg TriMix + 900 μg HIVACAT)
  Other Names: iHIVARNA-01.3
  Arms: 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA)

SUMMARY:
The main purpose of the study is to evaluate the safety and to establish the recommended dose of iHIVARNA-01 as a new therapeutic vaccine against HIV

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years of age
2. Voluntarily signed informed consent
3. Patient is male, or female with negative pregnancy test prior to enrolment
4. Patient has a proven HIV-1 infection (with positive antibodies against HIV-1 and a detectable plasma HIV-1 RNA before cART)
5. Patient must be on stable treatment with cART for at least 6 months (cART is defined as an antiretroviral regimen consisting of at least three registered antiretroviral agents)
6. Nadir CD4+ cell counts must be above or equal to 350 cells/μl (1 or 2 occasional determinations below 350 will be allowed)
7. Current CD4+ cell count must be at least 450 cells/μl
8. HIV-RNA must be below 50 copies/ mL for the last 6 months prior to inclusion, during at least two measurements (occasional so called 'blips' up to 50 copies/mL are permitted)

Exclusion Criteria:

1. Treatment with a non-cART regimen of antiretroviral agents prior to the start of cART;
2. History of a CDC class C event (see Appendix V);
3. Patient is female and has a positive pregnancy test or the wish of pregnancy:
4. Active opportunistic infection, or any active infection or malignancy within 30 days prior to screening visit;
5. Therapy with immunomodulatory agents, including cytokines (e.g. IL2) and gamma globulin, or cytostatic chemotherapy within 90 days prior to screening visit;
6. Use of anti-coagulant medication;
7. Use of any investigational drug during the 90 days prior to study entry;
8. Previous failure to antiretroviral and/or mutations conferring genotypic resistance to antiretroviral therapy EudraCT No. 2014-004591-32 33 Protocol version 1.1, dated 10 February 2015
9. Any other condition which, in the opinion of the investigator, may interfere with the evaluation of the study objectives.
10. Active hepatitis C virus or hepatitis B virus co-infection
11. Non-subtype B HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe García, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Bacelona, Barcelona, Spain

REFERENCES:
- [Derived] Leal L, Guardo AC, Moron-Lopez S, Salgado M, Mothe B, Heirman C, Pannus P, Vanham G, van den Ham HJ, Gruters R, Andeweg A, Van Meirvenne S, Pich J, Arnaiz JA, Gatell JM, Brander C, Thielemans K, Martinez-Picado J, Plana M, Garcia F; iHIVARNA consortium. Phase I clinical trial of an intranodally administered mRNA-based therapeutic vaccine against HIV-1 infection. AIDS. 2018 Nov 13;32(17):2533-2545. doi: 10.1097/QAD.0000000000002026. PMID 30289805

RESULTS

PARTICIPANT FLOW:
Groups:
- 100 μg TriMix mRNA (TriMix_100): Cohort 1 (control group) 3 patients will receive 100 μg of mRNA (i.e. 100 μg TriMix mRNA).If two or more of the three patients have a dose limiting toxicity (DLT), DSMB should be consulted and study will be terminated. If one or no patients have a dose limiting toxicity, three patients will be enrolled at the next dose level.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  TriMix_100: 100 μg of TriMix in
- 300 μg TriMix mRNA (TriMix_300): Cohort 2 (control group) 3 patients will receive 300 μg of mRNA (i.e. 100 μg TriMix mRNA).If two or more of the three patients have a DLT, DSMB should be consulted and study will be terminated. If one or no patients have a dose limiting toxicity, three patients will be enrolled at the next dose level.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  TriMix_300: 300 μg of TriMix in
- 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA): Cohort 3 (experimental group) 3 patients will receive 600 μg of mRNA (300 μg HIV mRNA + 300 μg TriMix mRNA). If two or more of the three patients have a DLT, DSMB should be consulted and study will be terminated. If one or no patients have a dose limiting toxicity, three patients will be enrolled at the next dose level.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA): 600 μg of mRNA (300 μg TriMix + 300 μg HIVACAT)
- 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA): Cohort 4 (experimental group) 3 patients will receive 900 μg of mRNA (i.e. 600 μg HIV mRNA and 300 μg TriMix mRNA). If two or more of the three first patients have a DLT, then additional three patients will be enrolled at the previous level dose (dose will be reduced to 600 μg of mRNA per vaccination). If one or no patients have a DLT, additional three patients will be enrolled at 900 μg dose level. If two or more of the six patients receiving 900 μg of mRNA have a DLT, then additional 3 patients will be enrolled at the previous level dose (dose will be reduced to 600 μg of mRNA per vaccination). If one or no patients of the six patients have a DLT, six patients will be enrolled at the next dose level.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA): 900 μg of mRNA (300 μg TriMix + 600 μg HIVACAT)
- 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA): Cohort 5 (experimental group) 6 patients will receive 1200 μg of mRNA (i.e. 900 μg HIV mRNA + 300 μg TriMix mRNA) in case one or no patients of the six patients at the previous dose level have a DLT.
  Each patient will receive 3 immunizations (at weeks 0, 2 and 4).
  1200μg mRNA (900 μg HIV mRNA+300 μg TriMix mRNA): 1200 μg of mRNA (300 μg TriMix + 900 μg HIVACAT)
Period: Overall Study
Arm/Group | 100 μg TriMix mRNA (TriMix_100) | 300 μg TriMix mRNA (TriMix_300) | 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) | 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) | 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA)
Started | 3 | 3 | 3 | 6 | 6
Completed | 3 | 3 | 3 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 100 μg TriMix mRNA (TriMix_100) | 300 μg TriMix mRNA (TriMix_300) | 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) | 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) | 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 6 | 6 | 21
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 48 [48 to 51] | 51 [48 to 51] | 45 [37 to 46] | 55 [53 to 57] | 47 [43 to 55] | 51 [48 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 0 | 5
  Male | 2 | 2 | 2 | 4 | 6 | 16
Region of Enrollment [Number; unit: participants]
  Spain | 3 | 3 | 3 | 6 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: Safety as measured by dose limiting toxicity (DLT), defined as:
  * Grade 3 or above local adverse event (pain, cutaneous reactions including induration)
  * Grade 3 or above systemic adverse event (temperature, chills, headache, nausea, vomiting, malaise, and myalgia)
  * Grade 3 or above other clinical or laboratory adverse event confirmed at examination or on repeat testing respectively
  * Any event attributable to vaccination leading to discontinuation of the immunisation regimen
Time Frame: week 24
Measure: Number; unit: participants
Arm/Group | 100 μg TriMix mRNA (TriMix_100) | 300 μg TriMix mRNA (TriMix_300) | 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) | 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) | 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6
participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Secondary Endpoint: Immunogenicty - Changes in the Magnitude of Total HIV-1-specific Immune Response Against IN Peptide Pools as Measured by ELISPOT at Baseline and Weeks 4, 6, 8 and 24 Measured by ELISPOT at Baseline and Weeks 4, 6, 8 and 24.
Description: Changes in the magnitude of total HIV-1-specific immune response against IN peptide pools as measured by ELISPOT at baseline and weeks 4, 6, 8 and 24 Results were considered positive if the number of SFC/106 cells in stimulated wells was two-fold higher than that in unstimulated control wells, and if there were at least 50 SFC/106 cells after background subtraction.
Time Frame: weeks 4, 6, 8 and 24
Measure: Median (Standard Error); unit: Spot forming cells per million of cells
Arm/Group | 100 μg TriMix mRNA (TriMix_100) | 300 μg TriMix mRNA (TriMix_300) | 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) | 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) | 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6
Spot forming cells per million of cells
  Week 4 (IN) | 54 (134) | 88 (88) | 140 (156) | -4 (76) | -106 (58)
  Week 6 (IN) | -38 (33) | 69 (69) | 37 (101) | -38 (126) | -28 (61)
  Week 8 (IN) | -25 (65) | 105 (105) | 256 (148) | 60 (78) | 173 (132)
  Week 24 (IN) | 3 (108) | 177 (148) | -32 (16) | -10 (75) | -21 (114)

3. Secondary Outcome: Secondary Endpoint: Immunogenicty - Changes in the Magnitude of Total HIV-1-specific Immune Response Against OUT Peptide Pools as Measured by ELISPOT at Abseline and Weeks 4, 6, 8 and 24 Measured by ELISPOT at Baseline and Weeks 4, 6, 8 and 24.
Description: Changes in the magnitude of total HIV-1-specific immune response against OUT peptide pools as measured by ELISPOT at abseline and weeks 4, 6, 8 and 24.
  Results were considered positive if the number of SFC/106 cells in stimulated wells was two-fold higher than that in unstimulated control wells, and if there were at least 50 SFC/106 cells after background subtraction.
Time Frame: weeks 4, 6, 8 and 24
Measure: Median (Standard Error); unit: Spot forming cells per million of cells
Arm/Group | 100 μg TriMix mRNA (TriMix_100) | 300 μg TriMix mRNA (TriMix_300) | 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) | 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) | 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6
Spot forming cells per million of cells
  Week 4 (OUT) | 327 (555) | 76 (191) | 379 (27) | 135 (383) | -357 (124)
  Week 6 (OUT) | -226 (176) | 203 (224) | 138 (168) | 10 (285) | 1 (73)
  Week 8 (OUT) | 16 (246) | -34 (300) | 377 (176) | 596 (593) | 17 (129)
  Week 24 (OUT) | 3 (226) | 375 (314) | 81 (50) | 100 (350) | -42 (124)

4. Secondary Outcome: Secondary End Point: Effect on Reservoir
Description: Changes from baseline in the intracelullar viral RNA copy number per million cells during and after the immunzation at week 4, 6, 8 and 24
Time Frame: weeks 4, 6, 8 and 24
Population: Baseline values were normalized to 1.0 for all groups. Subsequent measurements represent fold changes relative to baseline.
Measure: Mean (Standard Deviation); unit: Ratio to baseline
Arm/Group | 100 μg TriMix mRNA (TriMix_100) | 300 μg TriMix mRNA (TriMix_300) | 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) | 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) | 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA)
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6
Ratio to baseline
  baseline | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0)
  week 4 | 1.00631482 (0.1075206) | 1.19031378 (0.23113804) | 1.17119845 (0.42523104) | 1.1 (0.56388583) | 0.8 (0.46580374)
  week 6 | 0.69999513 (0.67071396) | 0.82859145 (0.38883214) | 0.66586182 (0.09336465) | 1.1 (0.32910834) | 1.5 (1.3519809)
  week 8 | 0.85170504 (0.59755696) | 0.81154264 (0.5543859) | 0.73222371 (0.40380891) | 1.1 (0.92490517) | 0.9 (0.26581174)
  week 24 | 1.83520809 (0.44289206) | 0.99741551 (0.12959672) | 0.58142711 (0.16635469) | 0.9 (0.3606482) | 1.0 (0.253664)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | 100 μg TriMix mRNA (TriMix_100) | 300 μg TriMix mRNA (TriMix_300) | 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) | 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) | 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/3 | 4/6 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 μg TriMix mRNA (TriMix_100) (N=3) | 300 μg TriMix mRNA (TriMix_300) (N=3) | 600μg mRNA (300 μg HIV mRNA+300 μg TriMix mRNA) (N=3) | 900μg mRNA (600 μg HIV mRNA+300 μg TriMix mRNA) (N=6) | 1200μg mRNA(900 μg HIV mRNA+300 μg TriMix mRNA) (N=6)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
haemotthoids (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nightmare (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
otitis extern (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
flu-like syndrome (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0)
rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — After vaccination
dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Dizziness because painful after vaccination
fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
urethritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
urinary tract infrection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
cold sore (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
mumps (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
There was an error in the study product, see: https://insights.ovid.com/pubmed?pmid=31490219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No